CLINICAL TRIAL: NCT03784053
Title: The Effect of Immersive Virtual Reality on Perceived Occupational Performance, Perceived Occupational Satisfaction, and Quality of Life of Older Adults
Brief Title: Virtual Reality and Occupational Performance, Satisfaction, and Quality of Life of Older Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of the Sciences in Philadelphia (Other)
Responsible Party: Principal Investigator, Sara Benham, Assistant Professor and Director of Doctoral Projects, University of the Sciences in Philadelphia
Other Study IDs: 1341686
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Aging
Keywords: Older adults; Virtual reality; Quality of life; Occupation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immersive virtual reality: Participants will receive eight 30-minute sessions of immersive virtual reality.
  Interventions: Other: Immersive virtual reality

INTERVENTIONS:
Other: Immersive virtual reality — At the start of every session, the participants' top five occupational problems will be reviewed, and a list of apps corresponding to the desired occupational problem will be offered through the immersive virtual reality device (Oculus Go). There will be eight 30-minute virtual reality sessions.

SUMMARY:
Older adult participants will complete eight immersive virtual reality (VR) sessions with the researcher, within five weeks (no more than two sessions per week may be scheduled). The screening process and assessment measures are not included in the five weeks of virtual reality. Sessions will consist of 30 minutes of use of the virtual reality goggles. During the virtual reality sessions, participants will select from a list of Oculus Go apps related to their self-identified occupational performance issues. Participants are expected to complete the session while seated with the VR set secured on their head.

DETAILED DESCRIPTION:
Virtual reality (VR) may promote engagement in meaningful daily activities that is tailored to the individual's skill level, need, and significance to their individual context. There is limited research on measurable changes in perceived meaningful daily activities after utilizing immersive VR, specifically with a head mounted display. Only in recent years have head-mounted displays become less expensive and more commercially available for research and patron purchase. At the low cost of $250, the device is within the reach of many older adult community centers for leisure and recreational use. The researchers will measure changes in occupational performance, occupational satisfaction, and quality of life for the older adult members of a community center, after eight immersive VR sessions. Sessions will consist of 30 minutes of use of the virtual reality goggles. During the virtual reality sessions, participants will select from a list of Oculus Go apps related to their self-identified occupational performance issues. Participants are expected to complete the session while seated with the VR set secured on their head.

ELIGIBILITY:
Inclusion Criteria:

1. Older adults aged 55+ that attend Journey's Way
2. Members need to attend least twice a week

Exclusion Criteria:

1. Score of 17 or less on the MoCA
2. A self-report a history of any of the following: Seizures, epilepsy, dizziness, vertigo, or motion sickness, any current contagious skin and eye conditions, experience sensitivity to light, have or use hearing aids, and a pacemaker and/or a defibrillator.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The aim is to recruit community-dwelling, healthy older adults from one community center. Subjects will be excluded if they receive a score of 17 or less on the MoCA because this score is associated with individuals with Alzheimer's Disease (Trzepacz, Hochstetler, Wang, Walker, & Saykin, 2015). The second exclusion, for safety purposes, is recommended by the Oculus Go user manual.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-21 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2020-01-14 (Estimated)

PRIMARY OUTCOMES:
The Canadian Occupational Therapy Performance Measure (COPM) | 10 minutes
  The COPM is a standardized outcome measure that identifies an individual's perceived occupational performance and occupational satisfaction and detects change in these areas over time. Through a semi-structured interview, individuals will identify their difficulties with self-care, leisure, and productivity (Law et al., 2005). The client is asked to rate the importance of each of the occupations to his/her life using a 10-point rating scale (1 to 10). Then, the client will rate the performance and satisfaction of the occupations on a 10-point rating scale (1 to 10). Then, the average performance satisfaction is calculated (1 to 10) and the average satisfaction is calculated (1 to 10). Higher scores indicate better outcomes.

SECONDARY OUTCOMES:
World Health Organization Quality of Life BREF (WHOQOL-BREF) | 10 minutes
  The WHOQOL-BREF is an assessment used to measure an individual's perceived quality of life. It has 26 items across the following four domains: physical health, psychological health, social relationships, and environment. Items are scored on a scale of 1 to 5 (a higher score is a more favorable outcome). Raw scores are calculated of each domain, and then scores may be transformed to scores ranging from 4 to 20 within each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Benham, OTD, OTR/L, Principal Investigator — University of the Sciences
Locations (1):
- Journey's Way, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Law, M., Baptiste, S., Carswell, A., McColl, M., Polatajko, H., & Pollock, N. (2005). Canadian occupational performance measure (4th ed.). Ottawa, Ont.: Canadian Association of Occupational Therapists.
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Trzepacz PT, Hochstetler H, Wang S, Walker B, Saykin AJ; Alzheimer's Disease Neuroimaging Initiative. Relationship between the Montreal Cognitive Assessment and Mini-mental State Examination for assessment of mild cognitive impairment in older adults. BMC Geriatr. 2015 Sep 7;15:107. doi: 10.1186/s12877-015-0103-3. PMID 26346644